CLINICAL TRIAL: NCT01971086
Title: Treatment With Rhinospray Plus of Patients With Acute Rhinitis in the Everyday Curative Routine in Hungary
Brief Title: Treatment With Rhinospray Plus in Patients With Acute Rhinitis in the Everyday Curative Routine in Hungary
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 40.56
Record Dates: First submitted 2013-10-14; First posted 2013-10-29 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- acute rhinitis

SUMMARY:
Multi-centre, open-label, prospective, uncontrolled, single-arm, non-interventional study (NIS) with objective to collect and evaluate data concerning treatment with Rhinospray Plus in everyday curative routine treatment of acute rhinitis

DETAILED DESCRIPTION:
Study Design:

open, observational, single-arm, uncontrolled

ELIGIBILITY:
Inclusion criteria:

1. Patients who (or in case of 6-18 years old whose legal representative) have signed the Informed Consent
2. Male and female ambulatory outpatients being seen in a participating physicians office for routine care
3. Patients with a clinical diagnosis of Rhinitis acuta
4. Patient having the cognitive and functional abilities for answering the symptom specific questions
5. Patients having expressed the willingness to participate in this observational study
6. Patients at and above the age of 6
7. Rhinospray Plus naive patients (patients who have not used Rhinospray Plus before)

Exclusion criteria:

1. Uncooperative patients based on physicians judgement
2. Patients with any conditions making the application of Rhinospray plus contraindicated
3. Patients currently enrolled in any clinical trial which requires a change in medication for their respiratory problems
4. Withdraw of Informed Consent
5. Pregnancy or breast-feeding as stated in the Summary of Product Characteristic (SmPC)
6. Patients with clinical diagnosis of allergic rhinitis

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adults and children at and above 6 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Hungary (4):
  - 40.56.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 40.56.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 40.56.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 40.56.36004 Boehringer Ingelheim Investigational Site, Budapest

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Rhinospray Plus: Patients with acute rhinitis treated with a maximum of 4 puffs per nostril a day of Rhinospray Plus nasal spray in a real life setting for up to 10 days.
Period: Overall Study
Arm/Group | Patients Treated With Rhinospray Plus
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients from the Treated Set (TS) which includes all patients who were documented to have taken at least one dose of the investigational treatment.
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (20.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 154

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in the Mean of the 3 Single Symptom Scores (Blocked Nose, Sneezing and Running Nose) at the Closing/Final Visit.
Description: Patients scored the symptoms (blocked nose, sneezing and running nose) on a 4-point rating scale with 0=absent, 1=mild, 2=moderate, 3=severe. The range of the mean score thus could be between 0 and 3. The change in the mean of the 3 single scores was calculated by the score at the final visit minus the score at baseline. Therefore, a negative change represents an improvement of the mean score.
Time Frame: Baseline and up to day 11
Population: Patients from the Full Analysis Set (FAS) which includes all patients in the TS who have analysable data in at least one efficacy endpoint.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
units on a scale | -2 [-3 to 0.7]

2. Primary Outcome: The Mean of the 2 Single Quality of Life Improvement Scores at the Closing/Final Visit for Daytime Activities and Quality of Sleep
Description: The mean score of the following two "quality of life improvement" questions at the final/closing visit was calculated: "How did Rhinospray plus improve the quality of your daytime activities?" and "How did Rhinospray Plus improve the quality of your sleep?". The scores range from 1=strongly to 4=no improvement. Thus also the range of the mean score is from 1 to 4.
Time Frame: up to day 11
Population: Patients from FAS
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
units on a scale | 1 [1 to 3]

3. Secondary Outcome: The Change From Baseline in the Single Symptoms Scores ( Blocked Nose, Sneezing and Running Nose) at the Closing/Final Visit
Description: Patients scored the single symptoms (blocked nose, sneezing and running nose) at the end of each treatment day on a 4-point rating scale with 0=absent, 1=mild, 2=moderate, 3=severe. The changes in the 3 single scores were calculated by the single score at the final visit minus the single score at baseline. Therefore, a negative change represents an improvement of the single scores.
Time Frame: Baseline and up to day 11
Population: Patients from FAS.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
units on a scale
  Blocked Nose | -3 [-3 to 1]
  Sneezing | -1 [-3 to 2]
  Running Nose | -2 [-3 to 1]

4. Secondary Outcome: The Single Score of Quality of Life Improvement at the Closing/Final Visit for Daytime Activities
Description: The following "quality of life improvement" question at the final/closing visit were answered by the patients: "How did Rhinospray plus improve the quality of your daytime activities?"
Time Frame: up to 11 days
Population: Patients from FAS
Measure: Number; unit: participants
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Strongly | 231
  Moderately | 61
  Weakly | 8
  No improvement | 0

5. Secondary Outcome: The Single Score of Quality of Life Improvement at the Closing/Final Visit for Quality of Sleep
Description: The following "quality of life improvement" question at the final/closing visit were answered by the patients: "How did Rhinospray plus improve the quality of your sleep?" and "How did Rhinospray Plus improve the quality of your sleep?".
Time Frame: Up to day 11
Population: Patients from FAS
Measure: Number; unit: participants
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Strongly | 236
  Moderately | 51
  Weakly | 5
  No improvement | 8

6. Secondary Outcome: Subjective Assessment of the Physicians of Overall Treatment Efficacy at the Closing/Final Visit.
Description: The efficacy of the treatment was rated by the physician at the closing/final visit for every patient.
Time Frame: up to day 11
Population: Patients from FAS.
Measure: Number; unit: participants
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Very good | 222
  Good | 70
  Fair | 8
  Poor | 0

7. Secondary Outcome: Subjective Assessment of the Patient of Overall Treatment Efficacy at the Closing/Final Visit.
Description: The efficacy of the treatment was rated by the patient at the closing/final visit.
Time Frame: up to day 11
Population: Patients from FAS
Measure: Number; unit: participants
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Very good | 212
  Good | 74
  Fair | 12
  Poor | 1
  Missing | 1

8. Secondary Outcome: Subjective Assessment of the Physicians of Overall Treatment Tolerability at the Closing/Final Visit.
Description: The tolerability of the treatment was rated by the physician at the closing/final visit for every patient.
Time Frame: up to day 11
Population: Patients from TS.
Measure: Number; unit: participants
Groups:
- Patients Treated With Rhinospray Plus: Patients with acute rhinitis treated with a maximum of 4 puffs a day of Rhinospray Plus nasal spray in a real life setting for up to 10 days.
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Very good | 236
  Good | 64
  Fair | 0
  Poor | 0

9. Secondary Outcome: Subjective Assessment of the Patient of Overall Treatment Tolerability at the Closing/Final Visit.
Description: The efficacy of the treatment was rated by the patient at the closing/final visit.
Time Frame: up to day 11
Population: Patients from TS
Measure: Number; unit: participants
Arm/Group | Patients Treated With Rhinospray Plus
Number analyzed (Participants) | 300
participants
  Very good | 230
  Good | 62
  Fair | 7
  Poor | 0
  Missing | 1

ADVERSE EVENTS:
Time Frame: up to 11 days
Arm/Group | Patients Treated With Rhinospray Plus
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.